CLINICAL TRIAL: NCT02796846
Title: The Association of CPAP Compliance and Nocturnal Hypoxemia in the Perioperative Period
Brief Title: The Association of CPAP Compliance Study
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Dr. Frances Chung, Staff Anesthesiologist, University Health Network, Toronto
Other Study IDs: Version date: October 6, 2017
Record Dates: First submitted 2016-06-07; First posted 2016-06-13 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: CPAP (continuous positive airway pressure); OSA (Obstructive sleep apnea)
MeSH Terms: conditions — Sleep Apnea, Obstructive; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CPAP prescription group: Patients with a CPAP prescription (both compliant and noncompliant)
- Without a CPAP prescription: Patients without a CPAP prescription to satisfy our primary goals/objectives.

SUMMARY:
The purpose of this study is to evaluate the pre and postoperative CPAP compliance rate in OSA surgical patients with or without a CPAP prescription. In this study, all diagnosed OSA patients with or without a CPAP prescription will be approached for informed consent to enroll in the study. Documented OSA is defined as an OSA diagnosis based on a previous laboratory or portable PSG, or on the prescription of CPAP for OSA. The patients with a CPAP prescription will be followed up to determine their compliance with CPAP and data will be collected to determine the O2 saturation. Those patients with diagnosed obstructive sleep apnea without a CPAP prescription will also be followed to objectively determine the severity of OSA which would indicate whether they do not require CPAP owing to their mild OSA or they in fact may require CPAP due to change in weight etc. Preoperative overnight oximetry will be performed on all the OSA patients at home before surgery. In the postoperative period, all patients will be followed up with a nocturnal oximetry in the first two post-operative nights of hospital stay. Postoperative compliance to CPAP will be evaluated and recorded in all the patients. The patients' charts will be reviewed for any postoperative complications. The clinical management of patient will be left to the discretion of the perioperative care team.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common sleep-related breathing disorder. CPAP is established to be the first line treatment for OSA patients with improvement in quality of life and significant reduction in the incidence of cardiovascular events. However, the evidence on the efficacy of CPAP in the perioperative period is largely lacking. A prospective cohort study conducted by Brar et al. found that despite the use of prescibed CPAP therapy, 18% of OSA patients became hypoxic on the night following surgery and they advocated postoperative oximetry monitoring in CPAP treated OSA surgical patients.

The investigators would like to determine the effect of CPAP compliance in reducing postoperative hypoxia and other complications in the surgical patients with OSA. The results from this study would provide valuable data on the rate of non-compliance to CPAP in the surgical patients with a history of diagnosed OSA and a CPAP prescription and the impact of non-compliance to CPAP on postoperative outcomes, especially oxygen saturation.

In this study, all diagnosed OSA surgical patients with or without a CPAP prescription will be approached for informed consent to enroll in the study. All study participants will be monitored for O2 desaturation by using wrist-watch pulse oximeter at home for one night preoperatively and first 3 nights post-operatively at the hospital.

The subjects enrolled will bring their own CPAP units (certified by the hospital engineering department as per hospital policy) and mask to the hospital. The OSA patients without a CPAP prescription will be followed up perioperatively to determine the severity of their OSA and to ascertain the rationale of no CPAP prescription.

Pre and post-operative CPAP usage data will be collected through interviewing the patient, chart review and monitoring recording in the smart CPAP device.

ELIGIBILITY:
Inclusion Criteria:

1. All adult surgical patients (>18 yr) with a diagnosis of OSA with or without a CPAP prescription.
2. Scheduled for a non-cardiac surgery (general surgery, orthopedics, urology, plastic surgery and spine) that is expected to require a postoperative hospital stay of more than one night.

Exclusion Criteria:

1. They are unwilling or unable to give informed consent to the study.
2. They are on supplemental oxygen preoperatively (daytime or nocturnal).
3. They are pregnant.
4. Surgery included tonsillectomy, septoplasty, uvuloplasty, pharyngoplasty, tracheostomy, or prolonged (> 48 hrs) postoperative mechanical ventilation of the lungs is anticipated. These procedures/interventions are likely to cure or at least modify the severity of OSA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult surgical patients (>18 yr) with a diagnosis of OSA with or without a CPAP prescription.
  Scheduled for a non-cardiac surgery (general surgery, orthopedics, urology, plastic surgery and spine) that is expected to require a postoperative hospital stay of more than one night.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2015-06; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
CPAP compliance | (average CPAP use ≥ 4hrs / night).
  CPAP compliance (average CPAP use ≥ 4hrs / night)

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kanagala R, Murali NS, Friedman PA, Ammash NM, Gersh BJ, Ballman KV, Shamsuzzaman AS, Somers VK. Obstructive sleep apnea and the recurrence of atrial fibrillation. Circulation. 2003 May 27;107(20):2589-94. doi: 10.1161/01.CIR.0000068337.25994.21. Epub 2003 May 12. PMID 12743002
- [Background] Parish JM, Somers VK. Obstructive sleep apnea and cardiovascular disease. Mayo Clin Proc. 2004 Aug;79(8):1036-46. doi: 10.4065/79.8.1036. PMID 15301332
- [Background] Chung F, Ward B, Ho J, Yuan H, Kayumov L, Shapiro C. Preoperative identification of sleep apnea risk in elective surgical patients, using the Berlin questionnaire. J Clin Anesth. 2007 Mar;19(2):130-4. doi: 10.1016/j.jclinane.2006.08.006. PMID 17379126
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Young T, Peppard PE, Gottlieb DJ. Epidemiology of obstructive sleep apnea: a population health perspective. Am J Respir Crit Care Med. 2002 May 1;165(9):1217-39. doi: 10.1164/rccm.2109080. PMID 11991871
- [Background] Singh M, Liao P, Kobah S, Wijeysundera DN, Shapiro C, Chung F. Proportion of surgical patients with undiagnosed obstructive sleep apnoea. Br J Anaesth. 2013 Apr;110(4):629-36. doi: 10.1093/bja/aes465. Epub 2012 Dec 19. PMID 23257990
- [Background] Keamy MF 3rd, Cadieux RJ, Kofke WA, Kales A. The occurrence of obstructive sleep apnea in a recovery room patient. Anesthesiology. 1987 Feb;66(2):232-4. doi: 10.1097/00000542-198702000-00023. No abstract available. PMID 3813086
- [Background] Lamarche Y, Martin R, Reiher J, Blaise G. The sleep apnoea syndrome and epidural morphine. Can Anaesth Soc J. 1986 Mar;33(2):231-3. doi: 10.1007/BF03010837. PMID 3697820
- [Background] Nishino T, Shirahata M, Yonezawa T, Honda Y. Comparison of changes in the hypoglossal and the phrenic nerve activity in response to increasing depth of anesthesia in cats. Anesthesiology. 1984 Jan;60(1):19-24. doi: 10.1097/00000542-198401000-00005. PMID 6691591
- [Background] Esclamado RM, Glenn MG, McCulloch TM, Cummings CW. Perioperative complications and risk factors in the surgical treatment of obstructive sleep apnea syndrome. Laryngoscope. 1989 Nov;99(11):1125-9. doi: 10.1288/00005537-198911000-00004. PMID 2530406
- [Background] Catley DM, Thornton C, Jordan C, Lehane JR, Royston D, Jones JG. Pronounced, episodic oxygen desaturation in the postoperative period: its association with ventilatory pattern and analgesic regimen. Anesthesiology. 1985 Jul;63(1):20-8. doi: 10.1097/00000542-198507000-00004. PMID 4014768
- [Background] Sollevi A, Lindahl SG. Hypoxic and hypercapnic ventilatory responses during isoflurane sedation and anaesthesia in women. Acta Anaesthesiol Scand. 1995 Oct;39(7):931-8. doi: 10.1111/j.1399-6576.1995.tb04200.x. PMID 8848894
- [Background] Chung F, Elsaid H. Screening for obstructive sleep apnea before surgery: why is it important? Curr Opin Anaesthesiol. 2009 Jun;22(3):405-11. doi: 10.1097/ACO.0b013e32832a96e2. PMID 19412094
- [Background] Chung F, Liao P, Yegneswaran B, Shapiro CM, Kang W. Postoperative changes in sleep-disordered breathing and sleep architecture in patients with obstructive sleep apnea. Anesthesiology. 2014 Feb;120(2):287-98. doi: 10.1097/ALN.0000000000000040. PMID 24158049
- [Background] Liao P, Yegneswaran B, Vairavanathan S, Zilberman P, Chung F. Postoperative complications in patients with obstructive sleep apnea: a retrospective matched cohort study. Can J Anaesth. 2009 Nov;56(11):819-28. doi: 10.1007/s12630-009-9190-y. PMID 19774431
- [Background] Gupta RM, Parvizi J, Hanssen AD, Gay PC. Postoperative complications in patients with obstructive sleep apnea syndrome undergoing hip or knee replacement: a case-control study. Mayo Clin Proc. 2001 Sep;76(9):897-905. doi: 10.4065/76.9.897. PMID 11560300
- [Background] Hwang D, Shakir N, Limann B, Sison C, Kalra S, Shulman L, Souza Ade C, Greenberg H. Association of sleep-disordered breathing with postoperative complications. Chest. 2008 May;133(5):1128-34. doi: 10.1378/chest.07-1488. Epub 2008 Mar 13. PMID 18339794
- [Background] Kaw R, Chung F, Pasupuleti V, Mehta J, Gay PC, Hernandez AV. Meta-analysis of the association between obstructive sleep apnoea and postoperative outcome. Br J Anaesth. 2012 Dec;109(6):897-906. doi: 10.1093/bja/aes308. Epub 2012 Sep 6. PMID 22956642
- [Background] Memtsoudis S, Liu SS, Ma Y, Chiu YL, Walz JM, Gaber-Baylis LK, Mazumdar M. Perioperative pulmonary outcomes in patients with sleep apnea after noncardiac surgery. Anesth Analg. 2011 Jan;112(1):113-21. doi: 10.1213/ANE.0b013e3182009abf. Epub 2010 Nov 16. PMID 21081775
- [Background] Mokhlesi B. Empiric postoperative autotitrating positive airway pressure therapy: generating evidence in the perioperative care of patients at risk for obstructive sleep apnea. Chest. 2013 Jul;144(1):5-7. doi: 10.1378/chest.13-0017. No abstract available. PMID 23880670
- [Background] Gilmartin GS, Tamisier R, Curley M, Weiss JW. Ventilatory, hemodynamic, sympathetic nervous system, and vascular reactivity changes after recurrent nocturnal sustained hypoxia in humans. Am J Physiol Heart Circ Physiol. 2008 Aug;295(2):H778-85. doi: 10.1152/ajpheart.00653.2007. Epub 2008 Jun 6. PMID 18539753
- [Background] Fletcher EC. Hypertension in patients with sleep apnoea, a combined effect? Thorax. 2000 Sep;55(9):726-8. doi: 10.1136/thorax.55.9.726. No abstract available. PMID 10950887
- [Background] Gami AS, Pressman G, Caples SM, Kanagala R, Gard JJ, Davison DE, Malouf JF, Ammash NM, Friedman PA, Somers VK. Association of atrial fibrillation and obstructive sleep apnea. Circulation. 2004 Jul 27;110(4):364-7. doi: 10.1161/01.CIR.0000136587.68725.8E. Epub 2004 Jul 12. PMID 15249509
- [Background] Rosenberg J, Ullstad T, Rasmussen J, Hjorne FP, Poulsen NJ, Goldman MD. Time course of postoperative hypoxaemia. Eur J Surg. 1994 Mar;160(3):137-43. PMID 8003566
- [Background] Squadrone V, Coha M, Cerutti E, Schellino MM, Biolino P, Occella P, Belloni G, Vilianis G, Fiore G, Cavallo F, Ranieri VM; Piedmont Intensive Care Units Network (PICUN). Continuous positive airway pressure for treatment of postoperative hypoxemia: a randomized controlled trial. JAMA. 2005 Feb 2;293(5):589-95. doi: 10.1001/jama.293.5.589. PMID 15687314
- [Background] Kaw R, Pasupuleti V, Walker E, Ramaswamy A, Foldvary-Schafer N. Postoperative complications in patients with obstructive sleep apnea. Chest. 2012 Feb;141(2):436-441. doi: 10.1378/chest.11-0283. Epub 2011 Aug 25. PMID 21868464
- [Background] Galatius-Jensen S, Hansen J, Rasmussen V, Bildsoe J, Therboe M, Rosenberg J. Nocturnal hypoxaemia after myocardial infarction: association with nocturnal myocardial ischaemia and arrhythmias. Br Heart J. 1994 Jul;72(1):23-30. doi: 10.1136/hrt.72.1.23. PMID 8068464
- [Background] Kehlet H, Rosenberg J. Late post-operative hypoxaemia and organ dysfunction. Eur J Anaesthesiol Suppl. 1995 May;10:31-4. PMID 7641641
- [Background] Lam B, Sam K, Mok WY, Cheung MT, Fong DY, Lam JC, Lam DC, Yam LY, Ip MS. Randomised study of three non-surgical treatments in mild to moderate obstructive sleep apnoea. Thorax. 2007 Apr;62(4):354-9. doi: 10.1136/thx.2006.063644. Epub 2006 Nov 22. PMID 17121868
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Weingarten TN, Flores AS, McKenzie JA, Nguyen LT, Robinson WB, Kinney TM, Siems BT, Wenzel PJ, Sarr MG, Marienau MS, Schroeder DR, Olson EJ, Morgenthaler TI, Warner DO, Sprung J. Obstructive sleep apnoea and perioperative complications in bariatric patients. Br J Anaesth. 2011 Jan;106(1):131-9. doi: 10.1093/bja/aeq290. Epub 2010 Oct 18. PMID 20959329
- [Background] Liao P, Luo Q, Elsaid H, Kang W, Shapiro CM, Chung F. Perioperative auto-titrated continuous positive airway pressure treatment in surgical patients with obstructive sleep apnea: a randomized controlled trial. Anesthesiology. 2013 Oct;119(4):837-47. doi: 10.1097/ALN.0b013e318297d89a. PMID 24195872
- [Background] Kohler M, Smith D, Tippett V, Stradling JR. Predictors of long-term compliance with continuous positive airway pressure. Thorax. 2010 Sep;65(9):829-32. doi: 10.1136/thx.2010.135848. PMID 20805182
- [Background] Mehta V, Subramanyam R, Shapiro CM, Chung F. Health effects of identifying patients with undiagnosed obstructive sleep apnea in the preoperative clinic: a follow-up study. Can J Anaesth. 2012 Jun;59(6):544-55. doi: 10.1007/s12630-012-9694-8. Epub 2012 Mar 30. PMID 22461134
- [Background] Kribbs NB, Pack AI, Kline LR, Smith PL, Schwartz AR, Schubert NM, Redline S, Henry JN, Getsy JE, Dinges DF. Objective measurement of patterns of nasal CPAP use by patients with obstructive sleep apnea. Am Rev Respir Dis. 1993 Apr;147(4):887-95. doi: 10.1164/ajrccm/147.4.887. PMID 8466125
- [Background] Reeves-Hoche MK, Meck R, Zwillich CW. Nasal CPAP: an objective evaluation of patient compliance. Am J Respir Crit Care Med. 1994 Jan;149(1):149-54. doi: 10.1164/ajrccm.149.1.8111574.
- [Background] O'Gorman SM, Gay PC, Morgenthaler TI. Does autotitrating positive airway pressure therapy improve postoperative outcome in patients at risk for obstructive sleep apnea syndrome? A randomized controlled clinical trial. Chest. 2013 Jul;144(1):72-78. doi: 10.1378/chest.12-0989. PMID 23287823
- [Background] Guralnick AS, Pant M, Minhaj M, Sweitzer BJ, Mokhlesi B. CPAP adherence in patients with newly diagnosed obstructive sleep apnea prior to elective surgery. J Clin Sleep Med. 2012 Oct 15;8(5):501-6. doi: 10.5664/jcsm.2140. PMID 23066360
- [Background] Sleep-related breathing disorders in adults: recommendations for syndrome definition and measurement techniques in clinical research. The Report of an American Academy of Sleep Medicine Task Force. Sleep. 1999 Aug 1;22(5):667-89. No abstract available. PMID 10450601
- [Background] Richard W, Kox D, den Herder C, Laman M, van Tinteren H, de Vries N. The role of sleep position in obstructive sleep apnea syndrome. Eur Arch Otorhinolaryngol. 2006 Oct;263(10):946-50. doi: 10.1007/s00405-006-0090-2. Epub 2006 Jun 27. PMID 16802139
- [Background] Charbonneau M, Marin JM, Olha A, Kimoff RJ, Levy RD, Cosio MG. Changes in obstructive sleep apnea characteristics through the night. Chest. 1994 Dec;106(6):1695-701. doi: 10.1378/chest.106.6.1695. PMID 7988186
- [Background] Weaver TE, Grunstein RR. Adherence to continuous positive airway pressure therapy: the challenge to effective treatment. Proc Am Thorac Soc. 2008 Feb 15;5(2):173-8. doi: 10.1513/pats.200708-119MG. PMID 18250209
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. Validation of the Berlin questionnaire and American Society of Anesthesiologists checklist as screening tools for obstructive sleep apnea in surgical patients. Anesthesiology. 2008 May;108(5):822-30. doi: 10.1097/ALN.0b013e31816d91b5. PMID 18431117
- [Background] Chung F, Yegneswaran B, Herrera F, Shenderey A, Shapiro CM. Patients with difficult intubation may need referral to sleep clinics. Anesth Analg. 2008 Sep;107(3):915-20. doi: 10.1213/ane.0b013e31817bd36f. PMID 18713905
- [Background] Chung F, Liao P, Sun Y, Amirshahi B, Fazel H, Shapiro CM, Elsaid H. Perioperative practical experiences in using a level 2 portable polysomnography. Sleep Breath. 2011 Sep;15(3):367-75. doi: 10.1007/s11325-010-0340-9. Epub 2010 Mar 16. PMID 20232260
- [Background] Chung F, Liao P, Elsaid H, Islam S, Shapiro CM, Sun Y. Oxygen desaturation index from nocturnal oximetry: a sensitive and specific tool to detect sleep-disordered breathing in surgical patients. Anesth Analg. 2012 May;114(5):993-1000. doi: 10.1213/ANE.0b013e318248f4f5. Epub 2012 Feb 24. PMID 22366847
- [Background] Ramakant Sharma ISB. CPAP for Obstructive Sleep Apnea in the Post-Operative Setting: An Oximetry Evaluation Study. J Sleep Disord Ther 2013;02.
- [Derived] Suen C, Wong J, Warsame K, Subramani Y, Panzarella T, Waseem R, Auckley D, Chaudhry R, Islam S, Chung F. Perioperative adherence to continuous positive airway pressure and its effect on postoperative nocturnal hypoxemia in obstructive sleep apnea patients: a prospective cohort study. BMC Anesthesiol. 2021 May 11;21(1):142. doi: 10.1186/s12871-021-01371-0. PMID 33975540